CLINICAL TRIAL: NCT02409069
Title: Influence of Non-invasive Neurostimulation (Transcutaneous Vagus Nerve Stimulation) on 1. the Noradrenergic Release in the Brain and 2. a Neuropsychological Memory Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Neurologie, Prof. dr. Kristl Vonck, University Hospital, Ghent
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EC/2014/0249
Record Dates: First submitted 2015-03-16; First posted 2015-04-06 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy; Cognitive Decline
Keywords: Transcutaneous vagus nerve stimulation; P300; Memory task
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transcutaneous vagus nerve stimulation (Nemos®, Cerbomed GmbH) (Experimental): Stimulation of the ramus auricularis of the vagus nerve (ear)
  Interventions: Device: Transcutaneous vagus nerve stimulation (Nemos®, Cerbomed GmbH)
- Sham stimulation (Nemos®, Cerbomed GmbH) (Sham Comparator): Stimulation of the earlobe
  Interventions: Device: Sham stimulation (Nemos®, Cerbomed GmbH)
- No stimulation (No Intervention): No stimulation

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation (Nemos®, Cerbomed GmbH)
  Arms: Transcutaneous vagus nerve stimulation (Nemos®, Cerbomed GmbH)
Device: Sham stimulation (Nemos®, Cerbomed GmbH)
  Arms: Sham stimulation (Nemos®, Cerbomed GmbH)

SUMMARY:
The goal of this study is to investigate the influence of transcutaneous vagus nerve stimulation 1. on the noradrenergic system in the brain and 2. on memory, in healthy volunteers.

Preclinical and clinical studies indicate that noradrenaline plays a role in the working mechanism of vagus nerve stimulation. This study will investigate if the effects of invasive vagus nerve stimulation can be replicated with transcutaneous vagus nerve stimulation.

The release of noradrenaline in the brain will be measured non-invasively by the P300 component of event-related potentials in the electro-encephalogram (EEG) via an auditory oddball paradigm.

Research to elucidate the working mechanism of non-invasive neurostimulation can help to identify subpopulations who will respond well to a treatment and can provide insights that could contribute to the optimalisation of the stimulation parameters, with as possible consequence a better clinical outcome.

Some studies indicate that stimulation of the vagus nerve can optimally influence memory, possibly via the noradrenergic system. This study will investigate if the effects of invasive vagus nerve stimulation on memory can be replicated with transcutaneous vagus nerve stimulation.

The influence of transcutaneous vagus nerve stimulation on memory will be measured via a neuropsychological memory task that investigates the ability to focus attention. The correlation between the performance on the memory task and the signal analysis of the auditory oddball task could give an indication about the underlying working mechanism of transcutaneous vagus nerve stimulation on memory.

This will be the first step to investigate whether transcutaneous vagus nerve stimulation can be used as innovative intervention for cognitive decline.

DETAILED DESCRIPTION:
First a sympathetic skin response (SSR) will be measured to investigate whether the SSR could be used as a method to measure the activity of the locus coeruleus non-invasively.

There are 3 conditions:

1. transcutaneous vagus nerve stimulation
2. sham stimulation
3. no stimulation

The conditions will be randomized.

In each condition the participant will do the oddball task and then the memory task. Between the conditions there is a wash-out period of 30 minutes. After completion of all 3 conditions and after a wash-out period of 30 minutes, the participant will do a final recognition task (part of the memory task in total).

During the oddball task EEG will be measured. An electro-cardiogram (ECG), electro-oculogram (EOG) and larynx electromyogram (EMG) will also be recorded for easy filtering of artefacts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 30 years
* Bachelor, Master or PhD students

Exclusion Criteria:

* Neurological or psychiatric disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Analysis of amplitude of P300 component of ERPs | 15 minutes
Performance on memory task as measured by number of correctly remembered words | 15 minutes

SECONDARY OUTCOMES:
Analysis of latency of P300 component of ERPs | 15 minutes
Performance on memory task as measured by number of correctly recognized words | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium